CLINICAL TRIAL: NCT06986499
Title: WSA Standard PMCF Study 2025
Brief Title: Standard Post Market Clinical Follow-up (PMCF) Study WSA 2025
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WSAUD A/S (Industry)
Collaborators: Hoerzentrum Oldenburg (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D00340960
Record Dates: First submitted 2025-05-12; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Hearing aid; Freiburger; Matrix Test; SSQ; IOI-HA
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of Study Device with Own devices (Other): within subject design: compare Widex SmartRIC MRRLD 440 to subjects' own hearing aids
  Interventions: Device: Hearing Aid Widex SmartRIC MRRLD 440; Device: Own hearing aid

INTERVENTIONS:
Device: Hearing Aid Widex SmartRIC MRRLD 440 — Receiver in Canal (RIC) hearing aid
Device: Own hearing aid — subjects' own hearing aids, any brand, any model

SUMMARY:
The purpose of the study is to follow-up on a released low-risk device as part of standard PMCF activities.

DETAILED DESCRIPTION:
This is a comparative study which is conducted monocentric at Hoerzentrum Oldenburg, Germany. The focus is to test a released hearing aid and compare this to the subject's own hearing aids with a minimum of 16 adult subjects with mild-to-moderate sensorineural hearing impairement. The subjects, all native German speakers, have 2 appointments of 1-2 hours including a fitting procedure with real-ear measurements and selected standard speech tests and undergo two 2-weeks home trials of the test hearing aid (with questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Sensorineural hearing loss, mild-to-moderately severe (Pure tone average of 500, 1000, 2000 and 4000 Hz <65).
* Hearing loss should fall within fitting range of study hearing aid
* Subjects should be experienced hearing aid users who have had and used hearing aids daily for at least 1 year.
* Air-Bone-Gap should be less or equal to 20 dB.
* Asymmetry between left and right ear should not exceed 20dB for frequencies in the range of 250Hz to 4kHz
* Healthy (outer and middle) ear
* Older than 18 years
* German is mother tongue
* Able to understand the instructions
* Willing to participate in laboratory tests and to wear the study HAs at home for 2 weeks
* Informed consent

Exclusion Criteria:

* Contraindication for HA treatment
* Fluctuating or rapidly progressing hearing loss
* "Central" hearing problems
* Limited mobility
* Limited dexterity (in handling the HA)
* Known psychological or cognitive problems
* Subjects must not show any injuries or a complete perforation of the ear drum. This must be clarified prior to the beginning of the study by means of otoscopy.
* Subjects should be in good overall medical condition (e.g., they shall not suffer from dementia) and should not use medical treatments that might affect study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Oldenburg Sentence Test | Estimated Time Frame 2 weeks (Test conducted at second lab session).
  The Oldenburg Sentence Test (OLSA) is an audiometric test for determining the speech recognition threshold in quiet and in noise. Sentences of the form name - verb - numeral - adjective - noun are used as speech material. The sequence of words is a random combination from an inventory of 50 words in total. The design of the test prevents memorization of the sentences, so the OLSA can be repeated as often as desired.

SECONDARY OUTCOMES:
Freiburger Monosyllabic Speech Test | Estimated Time Frame 2 weeks (Test conducted at second lab session).
  To investigate speech intelligibility (SI) performance for speech at 65dB in a quiet listening situation, the Freiburger monosyllabic speech test is used which is still the gold standard for Hearing Care Professionals (HCPs) in Germany.
Match-to-Target | Day 1 (Fitting procedure with real-ear measurements is done at first lab session)
  Investigate how close the study hearing aids fitted with the fitting software to NAL-NL2 Targets match the postulated targets, as measured in-situ with real-ear measurements
Speech, Spatial and Qualities of Hearing Questionnaire (SSQ) | 2 weeks
  A short form of the SSQ is used (SSQ 17, German version), to investigate speech perception, sound localisation, satisfaction and quality of hearing perceived in real-life. Responses are entered on a scale from 0 to 10, with 0 being the worst and 10 the best rating.
International Outcome Inventory for Hearing Aids (IOI-HA) | 2 weeks
  Investigate outcomes and effectiveness of hearing aid usage in real-life. Responses are entered on a 5-point scale with captions going from worst to best.
Satisfaction Questionnaire | 2 weeks
  Investigate satisfaction in real-life for different situations using proprietary questionnaire. Responses are entered on a 7 point likert scale with 1 signifying "Very dissatisfied" and 7 "very satisfied".
Basic User need questionnaire | 2 weeks
  Investigate ability to carry out different hearing aid functions of the test hearing aids in daily life using proprietary questionnaire. Subject can respond "Yes", "No" or "N.A.".

CONTACTS AND LOCATIONS:
Locations (1):
- Hörzentrum Oldenburg gGmbH, Oldenburg, Germany, Germany

IPD SHARING:
Plan to Share IPD: No